CLINICAL TRIAL: NCT01169792
Title: Association Between Genetic Polymorphisms of CYP2D6 and Outcomes in Breast Cancer Patients With Tamoxifen Treatment
Brief Title: Study of Cytochrome P450 Polymorphisms (CYP2D6, CYP3A4/5 and CYP2C19) in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Inje University (Other)
Other Study IDs: 4-2009-0483
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2009-10

CONDITIONS: Breast Neoplasms; Survival Analysis; Antineoplastic Agents; Therapeutic Uses
Keywords: Tamoxifen; Cytochrome P-450 CYP2D6; Polymorphism; Single nucleotide; Antineoplastic Agents, Hormonal
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples with DNA

GROUPS / COHORTS (1):
- Breast cancer patients: Breast cancer patients who underwent surgery with or without chemotherapy, endocrine therapy and/or radiation therapy. The patients are categorized according to the genetic polymorphisms or the activity score of the cytochrome P450 metabolism.
  Interventions: Drug: tamoxifen

INTERVENTIONS:
Drug: tamoxifen

SUMMARY:
The genetic polymorphisms of the cytochrome P450 may influence on the metabolism of tamoxifen.

The investigators want to

* evaluate the frequency or incidence of the genetic polymorphisms of cytochrome P450 subfamilies(CYP2D6, CYP3A4/5 and CYP2C19) in breast cancer patients, and
* analyze the association between the genetic polymorphisms of cytochrome P450 subfamilies and clinical outcomes in breast cancer patients treated by adjuvant tamoxifen therapy.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Breast cancer patients who underwent surgery

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors who underwent surgery at Severance hospital, Yonsei University Health System.
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
The frequency of the genetic polymorphisms of CYP2D6 in breast cancer patients
The frequency of the genetic polymorphisms of CYP3A4/5 in breast cancer patients
The frequency of the genetic polymorphisms of CYP2C19 in breast cancer patients

SECONDARY OUTCOMES:
The association between the genetic polymorphisms of CYP2D6 and outcomes in breast cancer patients with tamoxifen therapy
The association between the genetic polymorphisms of CYP3A4/5 and outcomes in breast cancer patients with tamoxifen therapy
The association between the genetic polymorphisms of CYP2C19 and outcomes in breast cancer patients with tamoxifen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Byeong-Woo Park, M.D.,ph.D., Study Chair — Department of Surgery and Brain Korea 21 Project for Medical Science, Yonsei University College of Medicine; Jae-Gook Shin, M.D.,ph.D., Study Chair — Department of Pharmacology and Pharmacogenomics Research Center, Inje University College of Medicine
Locations (2):
- South Korea (2):
  - Department of Pharmacology and Pharmacogenomics Research Center, Inje University College of Medicine, Jin-Gu, Busan
  - Department of Surgery, Yonsei University College of Medicine, Saedaemoon-gu, Seoul